CLINICAL TRIAL: NCT01207401
Title: Pain Control for Intrauterine Device Insertion: A Randomized Trial of 1% Lidocaine Paracervical Block
Brief Title: Paracervical Block Before Intrauterine Device (IUD) Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jessica Kiley, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00020958
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Results first posted 2013-06-10 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-05

CONDITIONS: Pain Control for Intrauterine Device Insertions
Keywords: intrauterine device; local anesthetic
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paracervical Block (Experimental)
  Interventions: Drug: Lidocaine
- No Paracervical Block (No Intervention)

INTERVENTIONS:
Drug: Lidocaine — 1% Lidocaine
  Arms: Paracervical Block

SUMMARY:
The purpose of this study is to evaluate if a paracervical block containing 1% lidocaine administered prior to IUD insertion reduces insertion pain. The hypothesis is that women receiving paracervical analgesia will experience less pain during IUD insertion than those who do not receive such analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 -50 years
* A negative urine pregnancy test and clinically unlikely to be pregnant
* Seeking an intrauterine device for any indication
* Willing and able to sign an informed consent in English

Exclusion Criteria:

* History of a prior IUD successful insertion
* Previous failed insertion of an IUD
* Known copper allergy
* Known levonorgestrel allergy
* Known lidocaine allergy
* Current cervicitis
* Pelvic Inflammatory Disease (PID) within 3 months
* Pregnancy within six weeks prior to IUD insertion
* Uterine anomaly or distortion of the uterine cavity
* Use of any other pain medication within 6 hours prior to IUD insertion
* Use of misoprostol within 24 hours prior to IUD insertion

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Kiley, MD MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Medical Faculty Foundation or Prentice Ambulatory Care Clinic, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: July 2010- February 2011, Northwestern Medical Faculty Foundation
Groups:
- Paracervical Block: IUD insertion after a 10 cc 1% Lidocaine administeration at 4 o'clock and 8 o'clock at the cervical-vaginal mucosa.
- No Paracervical Block: IUD insertion with no lidocaine injection
Period: Overall Study
Arm/Group | Paracervical Block | No Paracervical Block
Started | 26 | 24
Completed | 26 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paracervical Block | No Paracervical Block | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 24 | 50
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 31.9 (5.9) | 33.2 (6.2) | 32.6 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 50
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 24 | 50

OUTCOME MEASURES:

1. Primary Outcome: Median Visual Analogue Score Measuring Pain
Description: We asked participants to report their pain score on visual analogue scale (0mm=no pain and 100mm=worse pain possible) at the following time points:
  1. Speculum placement
  2. Tenaculum placement
  3. Paracervical block administration(if subject is in this arm)
  4. IUD insertion
  5. Five minutes post procedure
Time Frame: 1) Speculum placement 2) Tenaculum placement 3) Paracervical block administration(if subject is in this arm) 4) IUD insertion 5) Five minutes post procedure
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Paracervical Block | No Paracervical Block
Number analyzed (Participants) | 26 | 24
units on a scale
  1) Speculum Placement | 12 (13.1) [0 to 55] | 8.5 (12.9) [1 to 52]
  2) Tenaculum Placement | 12 (21.8) [0 to 98] | 28 (16.2) [0 to 57]
  3) Paracervical Block administration | 40 (29.3) [2 to 94] | NA [NA to NA] — VAS not administered because Group did not receive paracervical block
  4) IUD insertion | 24 (35.0) [0 to 99] | 62 (27.5) [2 to 89]
  5) 5 minutes post procedure | 12 (25.7) [0 to 97] | 17 (18.4) [1 to 66]

ADVERSE EVENTS:
Arm/Group | Paracervical Block | No Paracervical Block
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes